CLINICAL TRIAL: NCT00745927
Title: Application of CO2 Insufflations in Colonoscopy Examination-A Single-blinded Randomized Trial
Brief Title: Application of CO2 Insufflations in Colonoscopy Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 200802031R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Neoplasm; Colorectal Cancer
Keywords: Colorectal neoplasm; Colorectal cancer; Screening colonoscopy; CO2 insufflations; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Room air insufflations (No Intervention): Room air will be used for insufflations during colonoscopy
- CO2 insufflations (Active Comparator): CO2 will be used for insufflations during colonoscopy
  Interventions: Other: CO2 insufflations

INTERVENTIONS:
Other: CO2 insufflations — CO2 insufflations during whole procedure of colonoscopy
  Arms: CO2 insufflations

SUMMARY:
It has been reported that carbon dioxide (CO2) insufflation can reduce patient pain and abdominal discomfort during and after colonoscopy. Its safety and efficacy during colonoscopy even under sedation has been already assessed in some earlier trials. Air insufflation is still the standard method, however, because of a lack of suitable equipment and continued technical improvement in colonoscopy.

In laparoscopic surgery, CO2 insufflation is widely applied and safely used with the patient under general anesthesia. CO2 insufflation is also applied for CT colonography for reduction of discomfort during or after procedure.2 During endoscopic procedure for colorectal neoplasia resection, however, long procedural time may increase not only the degree of discomfort during and after the procedure but also the risk of perforation. In addition to laparoscopic surgery, CO2 insufflation has also been applied to other endoscopic procedures. Saito et al reported the application of CO2 insufflation in Endoscopic submucosal dissection (ESD) of colorectal neoplasia in a prospective study in which their average procedural time using CO2 insufflation was 90 minutes under conscious sedation with average of 5.6 mg of midazolam. When compared with control group using room air, statistically negligible difference of pCO2 was observed with significant difference in abdominal discomfort.6 Screening colonoscopy, which can be completed within 15 minutes if no lesion being detected, requires high screenee satisfaction so as to improve patient compliance. In the setting of colonoscopy after positive FOBT, the attendance rate for secondary colonoscopy was around 60 to 70 % according to the data demonstrated in previous RCT and population-based studies. With application of CO2 insufflation, further improvement of patient compliance can be anticipated.

This study aims to investigate whether use of CO2 insufflations can reduce examinee discomfort in comparison with air.

DETAILED DESCRIPTION:
* Setting: Screening colonoscopy or secondary colonoscopy after positive FOBT performed in endoscopic unit of a single university hospital
* Study design: Single blinded randomized trial
* Randomization process: sealed envelope
* Study subjects:

Inclusion criteria: Subjects who receive Screening colonoscopy or secondary colonoscopy Exclusion criteria: subjects who have COPD or cardiovascular diseases

* Study duration: June 2008 to November 2012
* Post-colonoscopy discomfort will be measured and obtained from the screenee at several time points using visual analogue pain scoring system:

  * Immediately after colonoscopy for non-sedated patients, immediately after awaken from sedation for sedated patients
  * 2 hrs after colonoscopy
  * 8-12 hours after colonoscopy
* Statistical analysis:

  * Sample size estimation: according to our previous unpublished data using air insufflations at colonoscopy, mean pain score was 3 and standard deviation was 2.38. Assuming 15% difference of discomfort, sample size up to 171 are required for each group (CO2 vs. air, sedated and non-sedated) in this study. (2 sided test, α=0.05, power=80%)
  * Student t-test for pain score comparison
  * Ancillary analysis: pCO2, sedation drug dosage, and procedural time in both groups. For TCCO2 comparison, ANOVA for repeated measurement will be used. For variables not normally distributed, Wilcoxon rank sum test wall be used as a supplementary analysis.
  * SAS statistical program, version 9.0 (SAS institute Inc., Cary, NC) will be used for all statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Subjects who receive Screening colonoscopy or secondary colonoscopy

Exclusion Criteria:

* Subjects who have COPD or cardiovascular diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Degree of abdominal discomfort during and after colonoscopy | 0, 2, 8-10 hr

SECONDARY OUTCOMES:
Number of neoplasm detected | At the time of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Po Wang, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan